CLINICAL TRIAL: NCT06597188
Title: Comparison of Transcatheter Aortic Valve Replacement With Surgical Aortic Valve Replacecment: A Prospective, Multicenter, International, Randomized Controlled, Non-inferiority Study for Bicuspid Aortic Valve Stenosis (PROMIS-BAV)
Brief Title: TAVR vs. SAVR Study of VitaFlow Liberty® for Severe BAV Stenosis
Acronym: PROMIS-BAV
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai MicroPort CardioFlow Medtech Co., Ltd. (Industry)
Collaborators: West China Hospital (Other); The First Affiliated Hospital of Anhui Medical University (Other); Zhejiang University (Other); Qilu Hospital of Shandong University (Other); People's Hospital of Xinjiang Uygur Autonomous Region (Other); Provincial Hospital of fuzhou University (Unknown); Yanan Hospital of Kunming City (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PROMIS-BAV-2024
Record Dates: First submitted 2024-09-10; First posted 2024-09-19 (Actual); Last update posted 2025-09-16 (Actual); Status verified 2025-09

CONDITIONS: Aortic Stenosis; Bicuspid Aortic Valve (BAV)
Keywords: Aortic stenosis; Bicuspid Aortic Valve (BAV); TAVR; SAVR
MeSH Terms: conditions — Aortic Valve Stenosis; Bicuspid Aortic Valve Disease

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- TAVR group (Experimental): TAVR with the study device will be performed in the TAVR group
  Interventions: Device: VitaFlow Liberty
- SAVR group (Active Comparator): SAVR with a commercially available surgical bioprosthetic valve will be performed in the control group
  Interventions: Device: Commercially available surgical bioprosthetic valve

INTERVENTIONS:
Device: VitaFlow Liberty — All subjects randomized to the TAVR group will receive transcatheter aortic valve replacement (TAVR) with the study device of VitaFlow Liberty
  Arms: TAVR group
Device: Commercially available surgical bioprosthetic valve — All subjects randomized to the SAVR group will receive surgical aortic valve replacement (SAVR) with the control device of a commercially available surgical bioprosthetic valve.
  Arms: SAVR group

SUMMARY:
To evaluate the safety and effectiveness of the Transcatheter aortic valve and retrievable delivery system (VitaFlow Liberty®) for the treatment of severe bicuspid aortic valve (BAV) stenosis.

DETAILED DESCRIPTION:
Transcatheter aortic valve replacement (TAVR) has emerged as the first-line treatment for symptomatic severe AS currently, while TAVR for bicuspid aortic valve (BAV) stenosis has not been well demonstrated in randomized controlled trials, thus more randomized controlled studies of TAVR vs. SAVR are still needed to provide strong evidence that TAVR treatment for patients with BAV stenosis has good safety and effectiveness.

This study is a prospective, international multicenter, randomized controlled, non-inferiority clinical study, in which the study device (VitaFlow Liberty®) for TAVR is to be demonstrated as non-inferior to the control device (a commercially available surgical bioprosthetic valve) for SAVR in terms of the incidence of composite endpoint events (all-cause mortality, all strokes and re-hospitalizations) at 12 months postoperatively.

In this study, 452 eligible subjects will be randomly assigned to the study group (n=226) or the control group (n=226) in a 1:1 ratio. The subjects in study group will be treated with the TAVR surgery using the study device (VitaFlow Liberty®) , while the subjects in control group will be treated with the SAVR surgery using the control device (a commercially available surgical bioprosthetic valve), and clinical follow-ups will be performed at discharge (or 7 days after surgery), 30 days, 6 months, 12 months, and 2, 3, 4, 5 years after surgery, respectively.

ELIGIBILITY:
Inclusion Criteria:

1. Subject aged ≤ 75 years;
2. With symptomatic severe bicuspid aortic stenosis, defined as: peak flow velocity ≥ 4.0m/s, or mean trans-aortic pressure gradient ≥ 40mmHg, or aortic orifice area (AVA) ≤ 1.0cm2 (or AVA index ≤ 0.6cm2/m2) confirmed by echocardiography；
3. New York Heart Association (NYHA) cardiac function classification ≥ Class II;
4. With an intermediate or low risk of surgical procedures (STS score ≤8%) assessed by the local heart team;
5. Voluntarily participate in this study and sign the informed consent form.

Exclusion Criteria:

1. Known allergy or resistance to study device and control device components such as nitinol or contrast media;
2. Known contraindication or allergy to anticoagulant or antiplatelet medications and inability to tolerate the anticoagulant or antiplatelet therapy;
3. Known presence of active infective endocarditis or other active infection;
4. Known presence of severe vascular disease that precludes safe implantation of the prosthetic valve;
5. Ascending aorta width ≥50mm;
6. Previous prosthetic valve implantation (mechanical or bioprosthetic) in any heart place;
7. The aortic root anatomy not suitable for transcatheter aortic valve implantation confirmed by preoperative imaging (including aortic root calcification that influence the sufficient dilatation of the rposthetic valve);
8. Intracardiac mass, left ventricular or left atrial thrombus, vegetations confirmed by preoperative echocardiography;
9. Acute myocardial infarction (defined as Q-wave MI or non-Q-wave MI) within 30 days prior to surgery;
10. Invasive therapeutic cardiac surgery within 30 days prior to surgery (except for temporary pacemaker or implantable cardioverter-defibrillator implantation);
11. Clinically diagnosed stroke or TIA within 3 months prior to surgery;
12. Gastrointestinal bleeding requiring hospitalization or transfusion therapy or other clinically significant bleeding or coagulation disorders within 3 months prior to surgery, which preclude the required antiplatelet therapy in the study;
13. Comorbid with severe native coronary artery lesions that require revascularization therapy;
14. Comorbid with severe mitral or tricuspid regurgitation;
15. Comorbid with cardiogenic shock or hemodynamic instability requiring support from positive inotropic agents or mechanical ventilation or mechanical cardiac assistance;
16. Comorbid with severe left ventricular dysfunction (defined as left ventricular ejection fraction LVEF <20%);
17. Comorbid with end-stage renal diseases requiring chronic dialysis;
18. Comorbid with blood dyscrasias defined as leukopenia (white blood cell count < 3×109/L), thrombocytopenia (platelet count < 50×109/L), history of bleeding diathesis or coagulopathy, or hypercoagulable states;
19. Subjects corresponding to the criteria of a vulnerable population (including patients who are unable to fully understand all aspects of the study, patients lacking capacity in the informed consent procedure and patients with dementia and cognitive impairment);
20. Female subjects known to be pregnant or lactating;
21. Life expectancy is less than 12 months as assessed by the investigator;
22. Subject is participating in or planning to participate in other drug or device clinical studies within 12 months postoperatively;
23. Any other condition that, at the discretion of investigator or heart team, may preclude the subject's safe participation in the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 452 (Estimated)
Dates: Start 2025-09-08 (Actual); Primary Completion 2028-09-30 (Estimated); Study Completion 2032-09-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of composite endpoint events (all-cause mortality, all strokes, and re-hospitalizations [surgery, valve or heart failure related re-hospitalizations]) | 12 months postoperatively
  The composite endpoint event at 12 months postoperatively refers to all-cause mortality, all strokes, and re-hospitalizations related to procedure, valve or heart failure that occur within 12 months postoperatively.

SECONDARY OUTCOMES:
Device success rate | 30 days postoperatively
  Device success is defined as meeting all the following criteria:
  1. Correct positioning of a single prosthetic heart valve into the proper anatomical location;
  2. Successful access, delivery of the device, and retrieval of the delivery system;
  3. Freedom from mortality;
  4. Freedom from surgery or intervention related to the devicea or to a major vascular or access-related or cardiac structural complication;
  5. Intended performance of the valvec (mean gradient <20mmHg, peak velocity <3 m/s, Doppler velocity index ≥ 0.25, and less than moderate aortic regurgitation).
Prosthetic valve performance evaluation | 30 days, 6 months, 12 months, 2-5 years postoperatively
  The prosthetic valve performance will be evaluated independently by the corelab based on the echocardiography.
New York Heart Association grading assessment of cardiac function | Discharge, 30 days, 6 months, 12 months, 2-5 years postoperatively
  New York Heart Association (NYHA) grading system includes four gradings with higher grading means severer outcome.
Quality of life assessment (Kansas City Cardiomyopathy Questionnaire score) | 30 days, 6 months, 12 months postoperatively
  Kansas City Cardiomyopathy Questionnaire (KCCQ) score is ranged from 0 to 100 with higher score means better quality of life.
All-cause mortality | 30 days, 6 months, 12 months, 2-5 years postoperatively
  According to the VARC3 criteria, all-cause mortality includes cardiovascular mortality and non-cardiovascular mortality.
Incidence of all strokes | 30 days, 6 months, 12 months, 2 to 5 years postoperatively
  According to the VARC3 criteria, all strokes include ischemic strokes (including TIAs), hemorrhagic strokes, and unspecified strokes, as well as disabling and non-disabling strokes.
Incidence of myocardial infarction | Discharge, 30 days, 6 months, 12 months, 2-5 years postoperatively
  Myocardial infarction in this study is defined according to the VARC3 criteria.
Incidence of major adverse cardiovascular and cerebrovascular events (MACCE) | 30 days, 6 months, 12 months postoperatively
  MACCE includes all-cause mortality, myocardial infarction, all strokes, and reoperation due to valvular dysfunction, with each event defined according to the VARC3 criteria.
Incidence of life-threatening or disabling major bleeding | 30 days, 6 months, 12 months, 2-5 years postoperatively
  Life-threatening or disabling major bleeding is defined as types 3 and 4 bleeding according to the VARC3 criteria.
Incidence of acute kidney injury (AKI) | Discharge, 30 days postoperatively
  According to the VARC3 criteria, AKI is defined as stages 2-4 acute kidney injury.
Incidence of conduction disturbance and arrhythmias | 30 days, 6 months, 12 months, 2-5 years postoperatively
  Conduction disturbance and arrhythmias are defined according to the VARC3 criteria.
Incidence of permanent pacemaker implantation | 30 days, 6 months, 12 months, 2-5 years postoperatively
  Defined as the percentage of subjects with newly permanent pacemaker implantation occurring after surgery among all subjects enrolled in each group.
Incidence of serious vascular complications | 30 days, 6 months, 12 months postoperatively
  Serious vascular complications are defined according to the VARC3 criteria.
Incidence of other TAVR-related complications | Immediately, 30 days, 6 months, 12 months, 2-5 years postoperatively
  Other TAVR-related complications include: conversion to surgery, unplanned cardiopulmonary mechanical assistance, coronary artery occlusion requiring intervention, ventricular septal perforation, mitral valve damage or dysfunction, cardiac tamponade, endocarditis, valvular thrombosis, valvular dyslocation (displacement, embolization, false release), and reoperation due to valve dysfunction (including surgical or interventional therapy).
Incidence of Bioprosthetic valve dysfunction (BVD) | 12 months, 2-5 years postoperatively
  BVD includes structural valve deterioration (SVD), moderate and severe prosthesis-patient mismatch (PPM), moderate and severe paravalvular leak (PVL), thrombosis or endocarditis.
Moderate to severe structural valvular deterioration (HVD) | 12 months, 2-5 years postoperatively
  Moderate HVD is defined as an increase in mean transvalvular gradient ≥ 10mmHg resulting in mean gradient ≥ 20mmHgc with concomitant decrease in EOA ≥ 0.3cm2 or ≥ 25% and/or decrease in Doppler velocity index ≥ 0.1 or ≥ 20% compared with echocardiographic assessment performed 1-3 months post-procedure, OR new occurrence or increase of ≥ 1 graded of intraprosthetic AR resulting in ≥ moderate AR.
  Severe HVD is defined as an increase in mean transvalvular gradient ≥ 20mmHg resulting in mean gradient ≥ 30mmHgc with concomitant decrease in EOA ≥ 0.6cm2 or ≥50% and/or decrease in Doppler velocity index ≥0.2 or ≥40% compared with echocardiographic assessment performed 1-3 months post-procedure, OR new occurrence, or increase of ≥ 2 grades,d of intraprosthetic AR resulting in severe AR
Bioprosthetic valve dysfunction (BVF) | 12 months, 2-5 years postoperatively
  BVF is a composite endpoint, including severe HVD, aortic valve reintervention, and valve-related mortality (investigator assessment).
Re-hospitalization related to procedure, valve or heart failure | 30 days, 6 months, 12 months, 2-5 years postoperatively
  Re-hospitalization related to procedure, valve or heart failure is defined according to the VARC3 criteria.
Incidence of adverse events (AEs) | throughout the clinical study period
  An AE is an untoward medical occurrence during the course of the clinical study, regardless of whether or not related to the study device
Incidence of serious adverse events (SAEs) | throughout the clinical study period
  Serious adverse event (SAE) refers to any adverse event that occurs during the clinical study of a medical device that results in any of the following:
  1. Leads to death, or
  2. Leads to serious deterioration of the health conditions, including:
     Fatal disease or injury Permanent defect in the physical structure or physical function Requiring hospitalization or prolongation of hospital stay Any event which requires medical or surgical intervention to prevent persistent disability/incapacity
  3. Leads to fetal distress, fetal death or congenital abnormality or congenital defect, etc.
  Note: Planned hospitalizations due to pre-existing disease conditions, or events that do not result in significant deterioration in health status due to procedures required by the clinical study program are not considered SAEs.

CONTACTS AND LOCATIONS:
Overall Officials: Mao Chen, Professor, Principal Investigator — West China Hospital
Locations (1):
- WEST CHINA Hospital of Sichuan University, Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: No